CLINICAL TRIAL: NCT00361530
Title: Effect of 3-hydroxy-3-methylglutaryl-coenzyme A(HMG-CoA) Reductase Inhibitor Upon Carotid Intima-media Complex Thickness in the Post-ischemic Patients With Hyperlipidemia During the Prospective Study of J-STARS.
Brief Title: Carotid Intima-media Thickness in Japan Statin Treatment Against Recurrent Stroke(J-STARS Echo)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government); Hiroshima University (Other); National Cerebral and Cardiovascular Center, Japan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: J-STARS echo; C000000212 (Other: UMIN CTR)
Record Dates: First submitted 2006-08-07; First posted 2006-08-08 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Ischemic Stroke
Keywords: stroke; brain ischemia; cerebrovascular accident; statin; hydroxymethylglutaryl-CoA Reductase Inhibitors; cholesterol; hypercholesterolemia; hyperlipidemia; multicenter studies; prospective studies; endpoint determination; randomized controlled trials; recurrence; pravastatin; plaque; tunica intima; tunica media; ultrasonography; carotid arteries
MeSH Terms: conditions — Ischemic Stroke; Stroke; Brain Ischemia; Hypercholesterolemia; Hyperlipidemias; Recurrence; Plaque, Amyloid | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

ARMS (2):
- Pravastatin (Active Comparator): Patient has 10mg oral administration of Pravastatin per day. It starts within one month from their entry and continues every day until the end of the study or its endpoints.
  Interventions: Drug: Statin
- No intervention (No Intervention): Patient has no intervention.

INTERVENTIONS:
Drug: Statin
  Arms: Pravastatin

SUMMARY:
Carotid ultrasound can reveal the intima-media complex thickness(IMT), that has been reported to be a marker of atherosclerosis as well as a risk of cardiovascular events, and to be attenuated by 3-hydroxy-3-methylglutaryl-coenzyme A (HMG-CoA) reductase inhibitors (statins) . This substudy of J-STARS will observe the temporal profile of carotid IMT prospectively in the patients with prescription of pravastatin and the control.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke except for cardiogenic embolism, from 1 month to 3 years after onset
* Hyperlipidemia and total cholesterol level of 180-240mg/dl without the prescription of statin within previous 30 days
* Able to visit outpatient department
* Informed consent on the form.

Exclusion Criteria:

* Ischemic stroke of other determined cause according to the TOAST classification
* Ischemic heart disease and necessary to use statin
* Hemorrhagic disorders
* Platelet count <=100,000/ul within 3 months prior to study start
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST)>= 100IU/L within 3 months prior to study start
* Serum creatinine >=2.0mg/dl within 3 months prior to study start
* A scheduled operation
* The presence of malignant disorder
* Patients whom carotid ultrasound cannot examine because of neck tumor or torticollis
* Patients after carotid endarterectomy or radiation therapy to neck
* Patients whose carotid ultrasound cannot be examined because of neck tumor or torticollis
* Patients after carotid endarterectomy or radiation therapy to neck

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 854 (Actual)
Dates: Start 2004-03; Primary Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Intima-media complex thickness (IMT) of the common carotid artery (CCA) | until the last day of the next February after 5-year follow-up survey

SECONDARY OUTCOMES:
Plaque score, number of plaque, recurrent cerebrovascular events | until the last day of the next February after 5-year follow-up survey

CONTACTS AND LOCATIONS:
Overall Officials: Masayasu Matsumoto, MD, PhD, Principal Investigator — Hiroshima University Hospital
Locations (2):
- Japan (2):
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - National Cardiovascular Center (NCVC), Suita-shi, Osaka

REFERENCES:
- [Derived] Wada S, Koga M, Kagimura T, Toyoda K, Nagai Y, Aoki S, Nezu T, Hosomi N, Origasa H, Ohtsuki T, Maruyama H, Yasaka M, Kitagawa K, Uchiyama S, Minematsu K, Matsumoto M; Japan Statin Treatment Against Recurrent Stroke (J-STARS) Echo Study Collaborators. Long-term changes in carotid intima-media thickness according to baseline blood pressure level: J-STARS Echo study. J Neurol Sci. 2025 Jan 15;468:123342. doi: 10.1016/j.jns.2024.123342. Epub 2024 Dec 9. PMID 39673820
- [Derived] Wada S, Koga M, Minematsu K, Toyoda K, Suzuki R, Kagimura T, Nagai Y, Aoki S, Nezu T, Hosomi N, Origasa H, Ohtsuki T, Maruyama H, Yasaka M, Kitagawa K, Uchiyama S, Matsumoto M. Baseline Carotid Intima-Media Thickness and Stroke Recurrence During Secondary Prevention With Pravastatin. Stroke. 2019 Jun;50(6):1586-1589. doi: 10.1161/STROKEAHA.119.024968. Epub 2019 Apr 30. PMID 31035902
- [Derived] Koga M, Toyoda K, Minematsu K, Yasaka M, Nagai Y, Aoki S, Nezu T, Hosomi N, Kagimura T, Origasa H, Kamiyama K, Suzuki R, Ohtsuki T, Maruyama H, Kitagawa K, Uchiyama S, Matsumoto M; J-STARS Investigators. Long-Term Effect of Pravastatin on Carotid Intima-Media Complex Thickness: The J-STARS Echo Study (Japan Statin Treatment Against Recurrent Stroke). Stroke. 2018 Jan;49(1):107-113. doi: 10.1161/STROKEAHA.117.018387. Epub 2017 Nov 30. PMID 29191850
- See also: Related Info — http://jstars.umin.ne.jp